CLINICAL TRIAL: NCT03278054
Title: Effect of Different Instrumentation Technique on Outcome of Primary Non Surgical Endodontic Treatment
Brief Title: Effect of Different Instrumentation Technique on Endodontic Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: seema
Record Dates: First submitted 2017-06-26; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Apical Periodontitis
Keywords: apical periodontitis; hybrid; ProTaper; rotary
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual group (Active Comparator): Root Canal Treatment with hand instruments:Root canal treatment was done with instrumentation using manual K files.
  Interventions: Other: Root Canal Treatment with hand instruments
- ProTaper group (Active Comparator): Root canal treatment with Protaper instruments:Root canal treatment was done using ProTaper rotary files S1, S2, F1, and F2.
  Interventions: Other: Root canal treatment with Protaper instruments
- Hybrid group (Active Comparator): Root canal treatment with hybrid instrumentation:Root canal treatment was carried out using ProTaper and Hyflex CM files.
  Interventions: Other: Root canal treatment with hybrid instrumentation

INTERVENTIONS:
Other: Root Canal Treatment with hand instruments — Root canal treatment was performed with K files.
  Arms: Manual group
Other: Root canal treatment with Protaper instruments — Root canals were enlarged with S1 S2 F1F2 F2 Protaper instruments
  Arms: ProTaper group
Other: Root canal treatment with hybrid instrumentation — Root canal were enlarged with combination of a combination of ProTaper Universal instruments to shape the coronal and middle thirds and Hyflex CM to prepare the apical third
  Arms: Hybrid group

SUMMARY:
Aim: To evaluate and compare the outcome of primary endodontic treatment following use of different instrumentation techniques.

Materials and methods: Study subjects were recruited from the pool of patients referred for the non-surgical root canal treatment in the Department of Conservative Dentistry & Endodontics at PGIDS, Rohtak (Haryana).

The study population comprised of patients requiring primary root canal treatment following the diagnosis of pulpal necrosis with chronic apical periodontitis in mature mandibular first and second molars.

Subjects were allocated to one of the three study groups: manual instrumentation, ProTaper instrumentation and Hybrid instrumentation.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES

The present study has been designed with the following aims and objective:

* To evaluate the effect of manual / rotary/hybrid instrumentation techniques on success of primary non surgical root canal treatment in teeth with apical periodontitis.
* To assess the incidence of postoperative pain in teeth treated with and without rotary instrumentation.
* To compare manual, rotary and hybrid instrumentation techniques in terms of periapical healing in teeth with apical periodontitis.

METHODOLOGY

Prior to treatment a thorough clinical and radiological examination was carried out. A thorough history was taken from each patient. Prior informed consent was taken after explaining the procedure, risks and benefits.

Clinical procedure: A total of 90 patients (n=30 in each group) were included in the study. Mature mandibular permanent molar with diagnosis of apical periodontitis (as confirmed clinically & by periapical radiograph) were chosen for the study. Patients were randomly allocated into three groups :Group I- manual instrumentation, Group II -rotary instrumentation (ProTaper) and Group III -Rotary instrumentation (Hybrid ).

After administration of local anesthesia, rubber dam isolation of the involved tooth was done. Caries excavation was done and access cavity was prepared using carbide burs in high speed handpiece with copious irrigation.Debridement of the pulp chamber was done and all canal orifices were identified. Negotiation of canals was done. Working length was determined using root ZX apex locator and verified radiographically. Instrumentation was done as follows.

GROUP A: Manual instrumentation: Hand instrumentation with the stainless steel K files was performed using step back technique.

GROUP B: Rotary instrumentation (ProTaper files): The cleaning and shaping of the canals was completed in accordance with a crown down technique recommended by the manufacturer, using the following operative sequence. Canals were instrumented with ProTaper rotary instruments. Recapitulation was carried out with size 10 k file.

GROUP C: rotary instrumentation (Hybrid): Roots canals were shaped with a combination of two NiTi rotary systems: ProTaper Universal instruments were used to shape the coronal and middle thirds and Hyflex CM files to prepare the apical third.

After completion of canal instrumentation in all the groups, canals were irrigated with 5.0 mL of 17% ethylene-diamine-tetra acetic acid for 1 minute followed by a final irrigation with 5.0 mL of 5.25% sodium hypochlorite. Canals were then be dried with sterile paper points. A lentulo-spiral was used to fill all canals with a Calcium hydroxide paste and the access cavity to be restored with intermediate restorative material. The patient were recalled after 1 week. At the second appointment, the calcium hydroxide paste were removed by using circumferential filing with Hedstrom files and copious irrigation with 5.25% sodium hypochlorite followed by 5.0 mL of 17% ethylenediaminetetraacetic acid and a final rinse of 5.0 mL 5.25% sodium hypochlorite. Canals were dried with the help of absorbent paper points and obturated. After obturation, the cavity was permanently restored. Immediate post-operative radiograph was then taken using preset exposure parameters and processed manually.

FOLLOW UP

Follow up and clinical and radiographic examination was carried out at 3, 6, 9 & 12 month period.

Outcome variables

* The primary outcome variables observed for the study was long term clinical and radiographic success rates.
* The secondary outcome measure was the incidence of postoperative pain.

Radiographic success: Radiographic success (change in Periapical Index score) of the root canal therapy was drawn by comparing the pre-operative; 3 month, 6month, 9 month & 12-month follow up radiographs.

Clinical success: it was determined by

* Absence of inter appointment flare ups and pain.
* Absence of tenderness to palpation /percussion
* Absence of sinus or any associated soft tissue swelling.
* Tooth mobility of grade I or less.
* No deterioration in periodontal pocket depth.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to participate in the study.
* Age greater than 18 years.
* No history of antibiotic use prior to treatment.
* Mature permanent mandibular molar having apical periodontitis requiring primary root canal treatment.
* There must be a radiographic evidence of periapical radiolucency and a diagnosis of pulpal necrosis, as confirmed by negative response to cold and electrical tests; and absence of bleeding on entering the pulp chamber.

Exclusion Criteria:

* Root canal retreatment.
* Failure to obtain authorization from patients.
* The presence of a difficult canal anatomy, internal or external resorption and immature teeth.
* Accident or complication during treatment like calcified canals, inability to achieve apical patency in any canals.
* Immuno-compromised, diabetic, pregnant and hypertensive patients.
* Periodontally compromised teeth.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Radiographic success | till 12 month period
  Periapical radiolucency was graded as Periapical Index (PAI) and scores less than 3 were grded as success
Clinical success | 12 months
  Absence of pain tenderness sinus or swelling was graded as clinical success

SECONDARY OUTCOMES:
Pain intensity | every 24 hours for 7 days
  Pain intensity before and after treatment was recorded using 0-100 mm VAS scale

IPD SHARING:
Plan to Share IPD: No